CLINICAL TRIAL: NCT03756168
Title: Clinical Evaluation of the Safety and Efficacy of a 1060 nm Diode Laser for Non-invasive Fat Reduction of the Flanks
Brief Title: Clinical Evaluation of the Safety and Efficacy of a 1060 nm Diode Laser (Flanks)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0518
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Fat Atrophy
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All subjects (Experimental)
  Interventions: Device: 1060nm Diode laser

INTERVENTIONS:
Device: 1060nm Diode laser — All subjects received a single treatment with Venus Bliss' 1064 nm laser administered to the flanks
  Venus Bliss is a non-invasive medical aesthetic device designed for body contouring. The device contains four 1060 nm diode laser applicators which are 60x60 mm in size. It has a separate RF/PEMF applicator, but this was not used in this study. There is a belt included with the system to allow for the secure attachment of the applicators to the treatment area.

SUMMARY:
The objective of this clinical study is to assess the safety and efficacy of using a 1060 nm diode laser for non-invasive fat reduction of the flanks.

DETAILED DESCRIPTION:
Open-label, baseline-controlled, evaluator-blind, multi-center study evaluating a 1060 nm diode laser for non-invasive fat reduction of the flanks. The study will enroll up to 50 subjects requesting non-invasive lipolysis of the flanks. Each subject will receive a single study treatment. Subjects will be followed at six weeks and twelve weeks post-treatment. Twelve week outcome will be compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* able to read, understand and voluntarily provide written informed consent
* healthy male or female > 18 years of age seeking treatment for unwanted fat in the abdomen
* BMI score is less then 30
* agree to not making any major changes in their diet or lifestyle during the course of the study
* able and willing to comply with the treatment / follow up schedule and requirements
* women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrolment and for the duration of the study, have a negative urine pregnancy test baseline

Exclusion Criteria:

* pregnant in the last 3 months intending to become pregnant, postpartum or nursing in the last 6 months
* any previous liposuction / lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months
* history of immunosuppression / immune deficiency disorders including AIDS and HIV infection, or use of immunosuppressive medications, 6 month prior to and during the course of the study
* History of hyperlipidemia, diabetes, hepatitis, blood coagulopathy or excessive bleeding
* Use of antiplatelet medications (81 mg of acetylsalicylic acid daily is permitted), anticoagulants, thrombocytes or any-inflammatory medications within 2 weeks of treatment
* Having a history of skin cancer or any other cancer in the area to be treated, including presence of malignant or pre-malignant pigmented lesions
* Having a permanent implant in the treatment area such as a metal plate or injected chemical substance such as silicone pr parenteral gold therapy (gold sodium thiomalate)
* Use of medications, herbs or food supplements and vitamins known to induce photosensitivity to light exposure at the wavelength used history of photosensitivity disorder
* Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections
* Tattoos in the treatment area
* Poor quality skin (laxity)
* Abdominal wall, muscular abnormality or hernia on physical examination
* Unstable weight within the last 6 months (+ or - 3% weight change in the prior six months)
* Participation in another clinical study involving the same anatomical areas within the last 6 months
* History of keloid and hypertrophic scar formation or poor wound healing in the treatment area
* As per the investigators discretion any physician or mental condition which may make it unsafe for the subject to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilmer, MD, Principal Investigator — Skin and Laser Centre of Northern California; Jeffery Kenkel, MD, Principal Investigator — UT Southwestern
Locations (2):
- United States (2):
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - UT Southwestern Medical Centre, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kang A, Kislevitz M, Wamsley C, Barillas J, Hoopman J, Kenkel J, Kilmer S. Clinical evaluation of the safety and efficacy of a 1060 nm diode laser for non-invasive fat reduction of the flanks. J Cosmet Dermatol. 2023 Nov;22(11):3017-3025. doi: 10.1111/jocd.15954. Epub 2023 Aug 22. PMID 37608607

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: All subjects received a single treatment with Venus Bliss' 1064 nm laser administered to the flanks
  Venus Bliss is a non-invasive medical aesthetic device designed for body contouring. The device contains four 1060 nm diode laser applicators which are 60x60 mm in size. It has a separate RF/PEMF applicator, but this was not used in this study. There is a belt included with the system to allow for the secure attachment of the applicators to the treatment area.
Period: Overall Study
Arm/Group | All Subjects
Started | 30
Had at Least 1 Treatment | 29
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- All Subjects Treated: All subjects received a single treatment with Venus Bliss' 1064 nm laser administered to the flanks
  Venus Bliss is a non-invasive medical aesthetic device designed for body contouring. The device contains four 1060 nm diode laser applicators which are 60x60 mm in size. It has a separate RF/PEMF applicator, but this was not used in this study. There is a belt included with the system to allow for the secure attachment of the applicators to the treatment area.
Arm/Group | All Subjects Treated
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type criteria
  I: Always burns, never tans Pale/ivory skin, Blue eyes, blond/red hair Mod. to severe freckles
  II: Usually burns, min tanning Fair skin, Blue/green/hazel eyes, blonde/red hair Light to moderate freckles
  III: Mild burns, uniform tanning Creamy white/fair skin, hazel/light brown eyes Dark blonde to light brown hair Min freckling
  IV: Burns minimally, tans well Light brown/olive skin, Brown eyes&hair
  V: Very rarely burns, tans easily/rapidly Dark brown/black skin, eyes&hair
  VI: Never tans or burns Black skin&hair Brown/black eyes
  Participants
    I | 0
    II | 15
    III | 8
    IV | 4
    V | 1
    VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in the Percentage of Fat Thickness From Baseline to 12-weeks Post-treatment
Description: Change in the percentage of fat thickness of the adipose layer as measured by ultrasound at 12 weeks post-treatment as compared to baseline.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: percentage of body fat
Groups:
- All Subjects: All subjects received a single treatment with Venus Bliss' 1064 nm laser administered to the flanks.
  Venus Bliss is a non-invasive medical aesthetic device designed for body contouring. The device contains four 1060 nm diode laser applicators which are 60x60 mm in size. It has a separate RF/PEMF applicator, but this was not used in this study. There is a belt included with the system to allow for the secure attachment of the applicators to the treatment area.
Arm/Group | All Subjects
Number analyzed (Participants) | 27
percentage of body fat | -6.9 (1.4)

2. Secondary Outcome: Change in Abdominal Circumference From Baseline to 12 Weeks Post-treatment
Description: Change in the abdominal circumference at 12 weeks post-treatment as compared to baseline
Time Frame: Week 12
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | All Subjects
Number analyzed (Participants) | 27
centimeters | -0.87 (0.55)

3. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction with treatment at 12 weeks was assessed using the 5-point Likert subject satisfaction scale. 5 is very satisfied, while 1 is very unsatisfied
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 27
units on a scale | 3.3 (0.9)

4. Secondary Outcome: Treatment Pain
Description: Treatment pain assessed immediately post-treatment as measured using the Wong-Baker Faces Scale. Pain was measured on a scale from 0-10 (10 worst pain ever, to 0 no pain at all)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 29
score on a scale | 3.1 (2.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT03756168/Prot_SAP_000.pdf